CLINICAL TRIAL: NCT05783830
Title: A Phase 0, Open-label, Non-controlled Study to Evaluate the Pharmacokinetics of a Single Intravenous Microdose of ACD856 in Healthy Volunteers
Brief Title: Study Evaluating the Pharmacokinetics of a Single Microdose of ACD856
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AlzeCure Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2000C0-001
Record Dates: First submitted 2021-04-01; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Cognition Disorder; Alzheimer Disease
Keywords: Cognition Disorder; Alzheimer's Disease
MeSH Terms: conditions — Cognition Disorders; Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACD856 (Experimental)
  Interventions: Drug: ACD856

INTERVENTIONS:
Drug: ACD856 — IV injection 100 mcg

SUMMARY:
This is a Phase 0, open-label, non-controlled, single-centre study designed to evaluate the pharmacokinetics (PK) and safety and tolerability of a single, bolus intravenous (iv) injection of a microdose of ACD856 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged >18 and <65 years.
* Signed and dated informed consent prior to any study-mandated procedure
* Willing and able to comply with study requirements.
* BMI >18.0 and <30.0 kg/m^2
* Male subjects must be willing to use condom or be vasectomised or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of dosing until 3 months after dosing with the IMP.
* Clinically normal medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.

Exclusion Criteria:

* History of any clinically significant disease or disorder which may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Any planned major surgery within the duration of the study.
* Clinically relevant findings in laboratory parameters, ECG or vital signs at screening
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity
* Regular use of any prescribed or non-prescribed medication
* Planned treatment or treatment with another investigational drug within 3 months
* Current smokers or users of nicotine products.
* Positive screen for drugs of abuse or alcohol at screening
* History of alcohol abuse or excessive intake of alcohol
* Presence or history of drug abuse
* History of, or current use of, anabolic steroids.
* Excessive caffeine consumption
* Plasma donation within one month of screening or blood donation during the 3 months prior to screening.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-04-18 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration vs time curve from time zero extrapolated to infinity | 24 hours
  a pharmacokinetic measure of the amount of study medication present in the blood
AUC from time zero to time of last quantifiable analyte concentration | 96 hours
  a pharmacokinetic measure of the amount of study medication present in the blood
Half-life associated with terminal slope of a semi-logarithmic concentration-time curve | 24 hours
  a pharmacokinetic measure of the time it takes for the study drug to be eliminated from the blood
Total body clearance following iv administration | 24 hours
  a pharmacokinetic measure of the time it takes for the study drug to be eliminated from the blood
Volume of distribution following iv administration | 24 hours
  a theoretical estimate of how much of the study drug that the body may contain

SECONDARY OUTCOMES:
Number of subjects with adverse events | 5 days
  how many participants have reported a drug related advers event
Number of subjects with clinically significant changes in vital signs | 5 days
  how many participants have had any clinically significant changes in vital signs
Number of subjects with clinically significant changes in 12-lead electrocardiograms (ECGs) | 5 days
  how many participants have had study drug related changes to cardiac function
Number of subjects with clinically significant changes in haematology and clinical chemistry and/or urinalysis | 5 days
  how many participants have had study drug related changes in laboratory test analyses

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sandin, Study Director — AlzeCure Pharma
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson B, Bylund J, Halldin MM, Rother M, Rein-Hedin E, Onnestam K, Segerdahl M. ACD856, a novel positive allosteric modulator of Trk receptors, single ascending doses in healthy subjects: Safety and pharmacokinetics. Eur J Clin Pharmacol. 2024 May;80(5):717-727. doi: 10.1007/s00228-024-03645-1. Epub 2024 Feb 14. PMID 38353689